CLINICAL TRIAL: NCT02965469
Title: The Syndemic of Stress and Aging in an HIV-infected Population
Brief Title: Psychosocial Stress and Aging in HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00033537; 1R03AG048033-01A1 (NIH)
Record Dates: First submitted 2016-11-04; First posted 2016-11-16 (Estimated); Last update posted 2022-04-15 (Actual); Status verified 2018-07

CONDITIONS: HIV; Aging; Stress, Psychological; Frailty
MeSH Terms: conditions — Stress, Psychological; Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): Participants randomized to this arm will have no change to their usual care
- Cell phone app (Experimental): Participants randomized to this arm will use a stress reduction cell phone app called "Breathe2Relax" to assess feasibility and acceptability
  Interventions: Behavioral: Breathe2Relax

INTERVENTIONS:
Behavioral: Breathe2Relax — The app teaches diaphragmatic breathing and has audiovisual coaching
  Other Names: cell phone app
  Arms: Cell phone app

SUMMARY:
This study will begin to assess the association between perceived stress and enhanced aging in persons living with HIV (PLWH). The investigators suspect this relationship may be mediated by increased aging within the immune system and subsequent low-level inflammation that commonly leads to multiple illnesses and frailty as one ages. The findings from this study will identify potential diagnostic and therapeutic targets to improve the health of aging PLWH which could also apply to HIV-uninfected populations.

DETAILED DESCRIPTION:
While life expectancy has increased markedly for people living with HIV (PLWH), gains in expected years of life have come at a cost - earlier onset and greater frequency of age-associated comorbid conditions, such as osteoporosis, metabolic syndrome, and cardiovascular disease. Accumulated multi-morbidity is the likely cause of much higher than age-expected rates of frailty in PLWH. Perceived stress is prevalent in PLWH and, when present, associated with worse clinical outcomes, including poor engagement in HIV care, rapid progression to AIDS, and higher AIDS-related mortality. Stress is a well-documented risk factor for many illnesses that demonstrate early onset in PLWH, and perceived stress has been hypothesized to be a cause of aging itself. Nonetheless, the role of perceived stress in early-onset aging and age-related illness in PLWH is essentially unexplored. Investigating the interrelatedness of aging, perceived stress, and HIV may elucidate mechanism(s) that underlie a phenotype of premature aging and functional decline in HIV patients with implications for understanding fundamental mechanisms of stress and aging in HIV uninfected populations. The proposed randomized controlled study will estimate correlations between perceived stress and both aging and HIV-specific outcomes and will measure feasibility of a cell phone-delivered stress reduction intervention. Participants will complete structured interviews to measure cumulative life stress, perceived stress, intimate partner violence exposure (as a traumatic stressor), functional status, frailty, and potential covariates across the age spectrum in PLWH. Stress measures will be correlated with biomarkers known to be associated with functional decline in aging, HIV-uninfected populations. The findings from this exploratory R03, led by a New Investigator, will measure feasibility of mobile technology for stress reduction interventions and estimate correlations between perceived stress and markers of aging and HIV disease. The results will be used to determine sample sizes necessary to perform definitive studies to assess the link between perceived stress and a phenotype of premature aging, as well as interventional studies of stress modification to mitigate the onset of early multi-morbidity and functional decline. These findings can be applicable to both HIV-infected and HIV-uninfected populations.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive serostatus
* Wake Forest ID clinic patient for at least 12 months
* prescribed ART for at least 6 months
* English fluency (cell phone app and some interview tools are only available in English)
* consistent access to a smartphone

Exclusion Criteria:

* ART-naive
* unable to perform functional measures
* recent (within 30 days) acute illness requiring medical therapy or hospitalization
* immunosuppressive agents (e.g. > 20 mg/d prednisone or equivalent, chemotherapy, biologic immune-modulating agents) in the last 6 months
* cancer requiring treatment within 3 years (except for non-melanoma skin cancer)
* use of non-steroidal anti-inflammatory drugs more frequently than once per week within the last 30 days.

Criteria iii-vi are necessary because of their effects on biomarkers of aging

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-05; Primary Completion 2017-11-14 (Actual); Study Completion 2017-11-14 (Actual)

PRIMARY OUTCOMES:
Correlation of perceived stress with HIV virologic suppression | 12 weeks
  Measure perceived stress using the Perceived Stress Scale (PSS) and calculate the correlation with HIV viral load
Correlation of perceived stress with immune senescence | 12 weeks
  Measure perceived stress using the Perceived Stress Scale (PSS) and calculate the correlation with biomarkers of immune senescence, including IL-6, soluble CD-14, telomere length, and DNA methylation
Correlation of perceived stress with inflammation | 12 weeks
  Measure perceived stress using the Perceived Stress Scale (PSS) and calculate the correlation with biomarkers of inflammation (C-reactive protein, salivary cortisol)
Correlation of perceived stress with frailty phenotype | 12 weeks
  Measure perceived stress using the Perceived Stress Scale (PSS) and calculate the correlation with each participant's Fried Frailty Index score (comprised of 5 items, including weight loss, exhaustion, 4 meter walk time, physical activity, and grip strength).

SECONDARY OUTCOMES:
Feasibility of a stress-reduction cell phone app | 12 weeks
  This outcome will measure the accrual, adherence and retention of using a stress-reduction cell phone application in people aging with HIV through the randomized pilot study.
The effect of a cell phone app on stress-reduction | 12 weeks
  The study will collect preliminary data on the efficacy of a cell phone-based stress reduction intervention versus usual care for improving markers of inflammation and aging, as well as HIV-specific outcomes.
Acceptability of a stress-reduction cell phone app | 12 weeks
  An exit survey will measure the acceptability of using a stress-reduction cell phone application in people aging with HIV.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine R Schafer, MD, Principal Investigator — Associate Professor
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No